CLINICAL TRIAL: NCT04750226
Title: An Open-Label Extension of Studies M15-736 and M20-339 to Evaluate the Safety and Tolerability of 24-Hour Daily Exposure of ABBV-951 in Subjects With Advanced Parkinson's Disease
Brief Title: Study To Assess Adverse Events and Change in Disease Activity Of 24-hour Continuous Subcutaneous Infusion Of ABBV-951 In Adult Participants With Advanced Parkinson's Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20-098; 2019-004204-35 (EudraCT Number)
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease; PD; ABBV-951; Levodopa/Carbidopa (LD/CD); Levodopa Phosphate/Carbidopa Phosphate (LDP/CDP)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ABBV-951 (Experimental): Participants will receive ABBV-951 by continuous subcutaneous infusion (CSCI) for 96 weeks during the Primary Treatment Period and during the optional Extended Treatment Period.
  Interventions: Drug: ABBV-951

INTERVENTIONS:
Drug: ABBV-951 — Solution for continuous subcutaneous infusion (CSCI).
  Other Names: Foscarbidopa; Foslevodopa

SUMMARY:
Parkinson's disease (PD) is a neurological condition, which affects the brain. PD gets worse over time, but how quickly it progresses varies a lot from person to person. Some symptoms of PD are tremors, stiffness, and slowness of movement. This study will assess how safe and effective ABBV-951 is in adult participants with PD. Adverse events and change in disease activity is evaluated.

ABBV-951 is an investigational (unapproved) drug containing Levodopa Phosphate/Carbidopa Phosphate (LDP/CDP) given as an infusion under the skin for the treatment of Parkinson's Disease. Adult participants with advanced PD and who have completed M15-736 or M20-339 study will be enrolled. Approximately 130 participants will be enrolled in the study in approximately 60 sites in the United States and Australia.

Participants will receive continuous subcutaneous infusion (CSCI) (under the skin) of ABBV-951 for 96 weeks during the Primary Treatment Period and during the optional Extended Treatment Period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical and remote telephone assessments, blood tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Completion of the parent study, Study M15-736 or Study M20-339.

Exclusion Criteria:

- Participant considered by the investigator to be an unsuitable candidate to receive ABBV-951 for any reason.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Event (AEs) | Up to Week 96
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An SAE is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above.
Percentage of Participants with AEs of Special Interest (AESIs) | Up to Week 96
  AESIs are defined as AEs from "special situations," such as accidental or intentional overdose, medication error, occupational or accidental exposure, off-label use, drug abuse, drug misuse, or drug withdrawal, all which must be reported whether associated with an AE or not.
Percentage Of Participants With Numeric Grade Equal To Or Higher Than 5 On The Infusion Site Evaluation Scale | Up To Week 96
  The Infusion Site Evaluation Scale will be used to assess infusion sites. Infusion Site Evaluation Scale is an eight-point numeric scale used to assess irritation at the infusion site area (0 being "no evidence of irritation" and 7 being "strong reaction spreading beyond the test site").
Percentage Of Participants With Letter Grade Equal To Or Higher Than D On The Infusion Site Evaluation Scale | Up To Week 96
  The Infusion Site Evaluation Scale will be used to assess infusion sites. Infusion Site Evaluation Scale is an A to G letter grade scale, used to assess irritation at the infusion site area (A being "no finding" to G being "Small petechial erosions and/or scabs").
Change From Baseline in Suicidality as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up To Week 96
  C-SSRS is a systematically administered instrument designed to assess suicidal behavior and ideation, track and assess all suicidal events, and assess the lethality of attempts. Any participant who has suicidal behavior or suicidal ideation with plan since the last C-SSRS completed, will be evaluated immediately by the investigator.
Change From Baseline in Impulsive-Compulsive Disorders and related behaviors as assessed in Parkinson's Disease- Rating Scale (QUIP-RS) | Up To Week 96
  The QUIP-RS is a brief, self-completed or rater-administered rating scale to assess the severity of symptoms of impulse control disorders (ICDs) and related behaviors reported to occur in PD. The QUIP-RS uses a 5-point Likert scale that requires individuals to rate the severity of each symptom based on its frequency.
Change From Baseline in Cognitive Impairment as Assessed by the Mini-Mental State Examination (MMSE) | Up To Week 96
  Cognitive impairment is assessed by the Mini-Mental State Examination (MMSE). MMSE is a brief 30-point questionnaire, administered by a trained rater, that provides a quantitative measure of cognitive status in adults and is used widely to screen for cognitive impairment and to estimate the severity of cognitive impairment at a given point in time, to follow the course of changes in a patient over time, and to document response to treatment.
Number of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed. | Up to Week 96
  Number of participants with abnormal change in clinical laboratory test results like hematology will be assessed..
Number of Participants with Abnormal Change From Baseline in Vital Sign Measurements like Systolic and Diastolic Blood Pressure will be Assessed | Up to Week 96
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Change From Baseline in Electrocardiograms (ECGs) | Up to Week 96
  12-lead resting ECGs will be recorded. Parameters include RR interval, PR interval, QT interval, and QRS duration.

SECONDARY OUTCOMES:
Change From Baseline in Average Normalized "On" Time as Assessed by the Parkinson's Disease (PD) Diary | Up To Week 96
  Change in "On" time without dyskinesia or with non-troublesome dyskinesia as assessed by the PD diary.
Change From Baseline in Average Daily Normalized "Off" Time as Assessed by the PD Diary | Up To Week 96
  Change in average daily normalized "Off" Time (Hours) is assessed based on PD Diary.
Change From Baseline in PD Symptoms as Assessed by the MDS-UPDRS Tool Part I | Up To Week 96
  The MDS-UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD) with scores ranging from 0 to 236 with 236 representing the worst disability, and 0 representing no disability.
Change From Baseline in Motor Experiences of Daily Living | Up To Week 96
  Motor experiences of daily living is assessed by the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II. The MDS-UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD) with scores ranging from 0 to 236 with 236 representing the worst disability, and 0 representing no disability.
Change From Baseline in PD Symptoms as Assessed by the MDS-UPDRS Tool Part III | Up To Week 96
  The MDS-UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD) with scores ranging from 0 to 236 with 236 representing the worst disability, and 0 representing no disability.
Change From Baseline in PD Symptoms as Assessed by the MDS-UPDRS Tool Part IV | Up To Week 96
  The MDS-UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD) with scores ranging from 0 to 236 with 236 representing the worst disability, and 0 representing no disability.
Change From Baseline in PD Symptoms as Assessed by the MDS-UPDRS Tool Parts I-III | Up To Week 96
  The MDS-UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD) with scores ranging from 0 to 236 with 236 representing the worst disability, and 0 representing no disability.
Change From Baseline in Sleep Symptoms | Up To Week 96
  Sleep symptoms are assessed by the Parkinson's Disease Sleep Scale-2 (PDSS-2). The PDSS-2 consists of 15 questions that evaluate motor and non-motor symptoms at night and upon wakening, as well as disturbed sleep.
Change From Baseline in Quality Of Life as Assessed by the PD Questionnaire-39 item (PDQ-39) | Up To Week 96
  Quality of life is assessed by the PD Questionnaire-39 item (PDQ-39). PDQ-39 is a disease-specific instrument designed to measure aspects of health that are relevant to participants with PD, and which may not be included in general health status questionnaires. Each item is scored on a 5-point scale.
Change From Baseline in Health-related Quality of Life as Assessed by EQ-5D-5L | Up To Week 96
  Health-related quality of life is assessed by EQ-5D-5L. EQ-5D-5L is a standardized instrument that consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue-scale (EQ-VAS).
Percentage Of Participants With Early Morning "Off" Assessed by the PD Diary as Percentage of Participants with early morning "Off" Upon Waking Up | Up To Week 96
  Early morning "Off" status is assessed by the PD Diary as percentage of participants with early morning "Off" upon waking up.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (52):
- United States (47):
  - University of Alabama at Birmingham - Main /ID# 217814, Birmingham, Alabama
  - University of South Alabama /ID# 218467, Mobile, Alabama
  - Xenoscience, Inc /ID# 222515, Phoenix, Arizona
  - Muhammad Ali Parkinson Center /ID# 218609, Phoenix, Arizona
  - Movement Disorders Center of Arizona /ID# 218471, Scottsdale, Arizona
  - Neuro Pain Medical Center /ID# 217720, Fresno, California
  - Loma Linda University Medical /ID# 217724, Loma Linda, California
  - University of California, Los Angeles /ID# 218460, Los Angeles, California
  - SC3 Research Group - Pasadena /ID# 223018, Pasadena, California
  - University of California, San /ID# 218595, San Diego, California
  - Duplicate_Cedars-Sinai Medical Center-West Hollywood /ID# 218607, West Hollywood, California
  - University of Colorado Hospital /ID# 218486, Aurora, Colorado
  - Alpine Clinical Research Center /ID# 218461, Boulder, Colorado
  - Denver Neurological Research, LLC /ID# 217811, Denver, Colorado
  - CenExel Rocky Mountain Clinical Research, LLC /ID# 217731, Englewood, Colorado
  - Georgetown University Hospital /ID# 218599, Washington D.C., District of Columbia
  - Visionary Investigators Network - Miami /ID# 217726, Miami, Florida
  - Renstar Medical Research /ID# 217837, Ocala, Florida
  - Neurology Associates Ormond Beach /ID# 217800, Ormond Beach, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida /ID# 222679, Port Charlotte, Florida
  - University of South Florida- Neuroscience Institute /ID# 218481, Tampa, Florida
  - Premiere Research Institute - Palm Beach /ID# 218743, West Palm Beach, Florida
  - Rush University Medical Center /ID# 217807, Chicago, Illinois
  - University of Chicago Medical /ID# 218611, Chicago, Illinois
  - St Elizabeth's Medical Center - Brighton /ID# 223082, Brighton, Massachusetts
  - St. Luke's Hosp. of Kansas City /ID# 218604, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 217723, St Louis, Missouri
  - Global Neurosciences Institute /ID# 218472, Lawrenceville, New Jersey
  - Northwell Health /ID# 218600, Lake Success, New York
  - M3 Wake Research Inc. /ID# 218482, Raleigh, North Carolina
  - The Orthopedic Foundation /ID# 218608, New Albany, Ohio
  - The Movement Disorder Clinic of Oklahoma /ID# 218580, Tulsa, Oklahoma
  - Legacy Medical Group - Neurology /ID# 217804, Portland, Oregon
  - University of Pennsylvania /ID# 218605, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital /ID# 218594, Philadelphia, Pennsylvania
  - Prisma Health-Upstate /ID# 217803, Greenville, South Carolina
  - Coastal Neurology /ID# 222893, Port Royal, South Carolina
  - KCA Neurology - Franklin /ID# 222811, Franklin, Tennessee
  - Vanderbilt University Medical Center /ID# 217722, Nashville, Tennessee
  - St. David's Healthcare Partnership, L.P., LLP /ID# 248148, Austin, Texas
  - Houston Pulmonary Sleep and Allergy Associates /ID# 218473, Cypress, Texas
  - Texas Movement Disorder Specialists /ID# 218610, Georgetown, Texas
  - Baylor College of Medicine /ID# 217728, Houston, Texas
  - University of Utah Health Care /ID# 218597, Salt Lake City, Utah
  - Neurological Associates - Forest Ave /ID# 218458, Richmond, Virginia
  - Inland Northwest Research /ID# 222520, Spokane, Washington
  - Duplicate_Medical College of Wisconsin /ID# 217721, Milwaukee, Wisconsin
- Australia (5):
  - Liverpool Hospital /ID# 221693, Liverpool, New South Wales
  - Westmead Hospital /ID# 218418, Westmead, New South Wales
  - Gold coast University Hospital /ID# 221694, Southport, Queensland
  - Royal Adelaide Hospital /ID# 218417, Adelaide, South Australia
  - The Royal Melbourne Hospital /ID# 218419, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Soileau M, Kumar R, Parab A, Brion T, White K, Yan CH, Shah MB, Kukreja P, Facheris MF, Shewale A, Aldred J. Patients' experience with and perspectives on long-term use of continuous subcutaneous infusion of foslevodopa/foscarbidopa in Parkinson's disease. J Neurol. 2025 May 22;272(6):416. doi: 10.1007/s00415-025-13123-y. PMID 40402298